CLINICAL TRIAL: NCT01782885
Title: Comparison of Acetaminophen and Platelet-rich Plasma Therapy for the Treatment of Knee Osteoarthritis.
Brief Title: Comparison of Acetaminophen and PRP Therapy for Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Mario Alberto Simental Mendia, M Sc, Principal Investigator, M. Sc., Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BI13-001
Record Dates: First submitted 2013-01-30; First posted 2013-02-04 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Platelet-Rich Plasma; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Active Comparator): Patients from this arm will receive a dosis of acetaminophen (500 mg/8 hours) while PRP treatment lasts.
  Interventions: Drug: Acetaminophen
- Intra-articular injection of PRP (Experimental): Patients from this arm will receive 3 intra-articular knee injections of autologous platelet-rich plasma, one injection every two weeks
  Interventions: Procedure: Intra-articular injection of PRP

INTERVENTIONS:
Procedure: Intra-articular injection of PRP — Patients from this arm will receive 3 intra-articular knee injections of autologous platelet-rich plasma, one injection every two weeks (6 weeks total).
  Arms: Intra-articular injection of PRP
Drug: Acetaminophen — Patients from this arm will receive a dosis of acetaminophen (500 mg/8 hours) while PRP treatment lasts (6 weeks total).
  Arms: Acetaminophen

SUMMARY:
The purpose of this study is to test whether the platelet-rich plasma (PRP) intra-articular injection therapy is effective as an alternative treatment option in patients with mild knee osteoarthritis within a controlled randomized study compared to first line treatment acetaminophen. The investigators will evaluate patients outcome in level of pain, knee function and quality of life before the treatment and at 6, 12 and 24 weeks follow up.

The study will be complemented with in vitro experiments of human osteoarthritic cartilage explants culture (treated with PRP) for histological and gene expression assays.

PRP intra-articular injections therapy is effective in patients with mild knee osteoarthritis by modifying the biochemical joint environment and cartilage regeneration capability.

DETAILED DESCRIPTION:
This is a randomized controled study. Patients enroled in the study will be divided into two groups (calculated n=30 per group). One group will be treated with acetaminophen (500 mg/8 h) for 6 weeks, the experimental group will receive a total of 3 intra-articular injections of PRP, one injection every 2 weeks. The intake of any other analgesic or anti-inflammatory drug will be prohibited in patients from two groups.

For those who received the infiltrations, the procedure consist of a 27-mL venous blood sample in 6 vacutainer tubes with sodium citrate 0.109 M for each injection. Samples are gently agitated to ensure mixing the anticoagulant with the blood. An extra tube with anticoagulated EDTA blood is obtained for initial platelet count. Blood samples are centrifuged for 10 minutes at 1800 rpm to separate the erythrocyte layer. The upper plasma layer is carefully collected in a new sterile propylene tube trying not to remove the leukocyte layer. Plasma from all tubes is centrifuged again for 12 minutes at 3400 rpm to obtain a two-part plasma: the upper part consisting on platelet-poor plasma and lower part consisting of platelet-rich plasma (PRP). The platelet-poor plasma is discarded to obtain a final volume of 3 mL. This volume, consisting of PRP, is mixed carefully through pipetting to resuspend platelets and it was then transferred to a new sterile glass tube. An aliquot of the final PRP is sent to the laboratory for platelet count. All open handling sample procedures are performed within a high-efficiency particulate air-filtered laminar flow hood.

Application of injections is carry out after disinfection of skin in the knee joint area. After local anesthesia with lidocaine chlorohydrate, platelets are activated using 10% calcium gluconate solution and the liquid PRP is injected in a sterile condition using a 22 G needle. The needle is inserted using the superolateral approach in an angle of approximately 45°.

Patients from PRP group will be asked to flex and extend their knees immediately after injection so that PRP could distribute adequately across the joint space. After 5-10 minutes of observation the patients are sent home with written indications including to have relative rest 24 to 48 hours after the injection, the use of cold therapy for 15 minutes three times a day and 500 mg of acetaminophen in case of pain and inflammation.

The use of NSAIDs or any steroids is prohibited. All the patients will be evaluated before the beginning of their respective treatment and at 6, 12 and 24 weeks after. Three different scales are used to evaluate clinical outcome, the VAS (Visual Analog Scale) that scores pain level, the WOMAC (Western Ontario and McMaster Universities Arthritis Index) which assesses pain, articular stiffness and functional limitation, and the Spanish (México) version of the SF-12 (Short Form-12) for assessment of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Patients who haven't received steroids injection or medical treatment 1 month before the study
* Patients with knee osteoarthritis grade I and II (Kellgren-Lawrence scale)
* Indistinct gender
* Patients who accept to participate in the study with previous signed informed consent

Exclusion Criteria:

* Patients with knee osteoarthritis grade III and IV (Kellgren-Lawrence scale)
* Patients with prosthesis
* Pregnancy
* Patients with rheumatic diseases
* Patients with diabetes, hepatic diseases, coagulopathy, cardiovascular diseases, immunosuppression, infections
* Patients taking anticoagulants
* Patients with concentrations of hemoglobin under 11 g/dL and platelets under 150,000/uL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario A. Simental, MSc, Principal Investigator — Universidad Autónoma de Nuevo León, Facultad de Medicina; Felix Vilchez, PhD, Study Director — Universidad Autónoma de Nuevo León, Hospital Universitario Dr. José E. González; Herminia G Martínez, PhD, Study Director — Universidad Autónoma de Nuevo León, Facultad de Medicina
Locations (1):
- Hospital Universitario Dr. José E. González, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879
- [Background] Filardo G, Kon E, Pereira Ruiz MT, Vaccaro F, Guitaldi R, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma intra-articular injections for cartilage degeneration and osteoarthritis: single- versus double-spinning approach. Knee Surg Sports Traumatol Arthrosc. 2012 Oct;20(10):2082-91. doi: 10.1007/s00167-011-1837-x. Epub 2011 Dec 28. PMID 22203046
- [Background] van Buul GM, Koevoet WL, Kops N, Bos PK, Verhaar JA, Weinans H, Bernsen MR, van Osch GJ. Platelet-rich plasma releasate inhibits inflammatory processes in osteoarthritic chondrocytes. Am J Sports Med. 2011 Nov;39(11):2362-70. doi: 10.1177/0363546511419278. Epub 2011 Aug 19. PMID 21856929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with degenerative osteoarthritis were recruited from May 2013 to November 2015 in the Service of Orthopedics and Traumatology at the University Hospital "Dr. José Eleuterio González" of the Autonomous University of Nuevo León in Monterrey, México.
Pre-assignment Details: Only patients meeting inclusion criteria were assigned to a group (radiographic grade I and II osteoarthritis, mainly). Importantly, patients with previous surgical interventions, with concomitant diseases or with Hb values of <11 g/dL and platelet values of <150,000/µL were excluded prior to group assignment.
Groups:
- Acetaminophen: Patients from this arm will receive a dose of acetaminophen (500 mg/8 hours) during 6 weeks.
- Intra-articular Injection of PRP: Patients from this arm will receive 3 intra-articular knee injections of autologous platelet-rich plasma, one injection every two weeks (6 weeks of treatment).
Period: Overall Study
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Started | 36 | 39
Completed | 32 | 33
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Acetaminophen: Patients from this arm will receive a dosis of acetaminophen (500 mg/8 hours) during 6 weeks.
- Intra-articular Injection of PRP: Intra-articular injection of PRP: Patients from this arm will receive 3 intra-articular knee injections of autologous platelet-rich plasma, one injection every two weeks (6 weeks treatment).
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Intra-articular Injection of PRP | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.4) | 57.2 (8.1) | 56.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 12 | 11 | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.5 (3.8) | 32.2 (6.2) | 30.9 (5.0)
Grade of Osteoarthritis [Number; unit: participants] — Grade 0: No radiographic features of osteoarthritis, Grade I: Possible joint space narrowing and osteophyte formation, Grade II: Definite osteophyte formation with possible joint space narrowing, Grade III: Multiple osteophytes, definite joint space narrowing, sclerosis and possible bony deformity, Grade IV: Large osteophytes, marked joint space narrowing, severe sclerosis and definite bony deformity
  participants
    Kellgren-Lawrence Grade I | 12 | 11 | 23
    Kellgren-Lawrence Grade II | 20 | 22 | 42
Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: cm] — The visual analog scale (VAS) is a psychometric response scale which measures subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their current level of pain by indicating a position along a continuous line of 10 cm. Subject is asked: on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain imaginable, what you rate your current pain?
  cm | 5.9 (2.2) | 4.9 (2.4) | 5.4 (2.3)
Western Ontario and McMaster Universities Arthritis Index (WOMAC) [Mean (Standard Deviation); unit: units on a scale] — The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). A total WOMAC score is created by summing the items for all three subscales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  units on a scale | 35.5 (19.0) | 35.7 (19.5) | 35.6 (19.3)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) is a psychometric response scale which measures subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their current level of pain by indicating a position along a continuous line of 10 cm. Subject is asked: on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain imaginable, what you rate your current pain?
Time Frame: 0-24 weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
Centimeters
  VAS (0 weeks) | 5.9 (2.2) | 4.9 (2.4)
  VAS (6 weeks) | 3.8 (2.2) | 1.9 (1.6)
  VAS (12 weeks) | 4.1 (2.6) | 1.9 (2.0)
  VAS (24 weeks) | 3.7 (2.7) | 2.2 (2.1)

2. Other Pre Specified Outcome: Change in SF-12v2 Health Survey
Description: The Spanish (Mexico) version of the SF-12v2 Health Survey uses 12 questions to measure functional health and well-being from the patient's point of view. All 12 items from the survey can be summarized in two main domains (physical and mental health). Physical and Mental Health Composite Scores (PCS and MCS) are computed using the scores of 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Mental Component Summary | 50.8 (9.9) | 44.2 (11.8)
  Physical Component Summary | 37.7 (9.3) | 38.0 (8.0)

3. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: The WOMAC evaluation will be performed on patients who received the treatment at 0, 6, 12, 24 weeks after treatment is finished. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). A total WOMAC score is created by summing the items for all three subscales (score range 0-96). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Stiffness (0 weeks) | 3.0 (2.1) | 2.9 (2.0)
  Pain (0 weeks) | 8.0 (4.3) | 7.4 (4.0)
  Functional capacity (0 weeks) | 24.4 (13.7) | 25.3 (14.3)
  Total score (0 weeks) | 35.5 (19.0) | 35.7 (19.5)

4. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: as for outcome 3
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Stiffness (6 weeks) | 2.3 (1.8) | 1.1 (1.1)
  Pain (6 weeks) | 5.8 (2.9) | 3.1 (2.6)
  Functional capacity (6 weeks) | 18.2 (12.0) | 8.7 (8.0)
  Total score (6 weeks) | 26.2 (16.0) | 12.8 (11.0)

5. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Stiffness (12 weeks) | 2.2 (2.2) | 0.9 (1.3)
  Pain (12 weeks) | 5.7 (4.1) | 2.7 (2.4)
  Functional capacity (12 weeks) | 18.4 (13.1) | 8.1 (7.2)
  Total score (12 weeks) | 26.3 (17.8) | 12.0 (10.6)

6. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: as for outcome 3
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Stiffness (24 weeks) | 1.9 (1.9) | 0.8 (1.1)
  Pain (24 weeks) | 5.3 (3.9) | 2.9 (2.2)
  Functional capacity (24 weeks) | 16.7 (13.3) | 7.9 (7.7)
  Total score (24 weeks) | 23.5 (18.4) | 11.7 (10.0)

7. Other Pre Specified Outcome: Change in SF-12v2 Health Survey
Description: as for outcome 2
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Mental Component Summary | 49.8 (9.3) | 55.4 (8.7)
  Physical Component Summary | 41.1 (9.9) | 47.6 (7.9)

8. Other Pre Specified Outcome: Change in SF-12v2 Health Survey
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Mental Component Summary | 50.7 (8.7) | 55.9 (7.9)
  Physical Component Summary | 41.7 (8.5) | 48.8 (7.9)

9. Other Pre Specified Outcome: Change in SF-12v2 Health Survey
Description: as for outcome 2
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Number analyzed (Participants) | 32 | 33
units on a scale
  Mental Component Summary | 52.3 (7.2) | 54.3 (7.6)
  Physical Component Summary | 41.4 (7.4) | 49.9 (8.1)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All patients were asked and evaluated for possibles adverse events at time-points of evaluation. Specific attention was provided for PRP treated patients.
Arm/Group | Acetaminophen | Intra-articular Injection of PRP
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=32) | Intra-articular Injection of PRP (N=33)
Pain, inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) — Some patients showed mild pain and inflammation at the site of injection after they were treated with PRP. These symptoms prevailed for 2-3 days after injection with spontaneous resolution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes